CLINICAL TRIAL: NCT04711161
Title: Ph 1/1B Evaluation of the Safety, Pharmacokinetics and Efficacy of GRN-300, a Salt-inducible Kinase Inhibitor, Alone and in Combination With Paclitaxel, in Recurrent Ovarian, Primary Peritoneal, and Fallopian Tube Cancers.
Brief Title: First-in-Human Evaluation of GRN-300 in Subjects With Recurrent Ovarian, Primary Peritoneal, and Fallopian Tube Cancers.
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Business/Commercial Reasons
Sponsor: Green3Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRN300-001
Record Dates: First submitted 2020-12-24; First posted 2021-01-15 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Tumors
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; taxane

STUDY DESIGN:
Intervention Model Description: GRN-300 single-agent and in combination with paclitaxel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Phase 1a): Single Arm, Open Label (GRN-300 single-agent) (Experimental): Part 1 of the study will determine the safety of continuous twice a day oral dosing of GRN-300, with each cycle consisting of 28 days of treatment. The number of administered cycles will depend on the tolerability of each dose level and the severity and occurrence of side effects and DLTs. The maximal tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of GRN-300 as a single agent will be determined. The overall duration of Part 1 will be approximately 24-36 months, depending on the rate of enrollment and the number of subjects enrolled.
  Interventions: Drug: GRN-300
- Part 2 (Phase 1b): Single Arm, Open Label (GRN-300 plus paclitaxel) (Experimental): The study will determine the safety of continuous twice a day oral dosing of GRN-300, with each cycle consisting of 28 days of treatment, in combination with intravenously administered paclitaxel weekly x 3 during each 28-day cycle. The number of administered cycles will depend on the tolerability of each dose level and the severity and occurrence of side effects and DLTs. The maximal tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of GRN-300 in combination with paclitaxel will be determined. The overall duration of Part 2 will be approximately 12-18 months, depending on the rate of enrollment and the number of subjects enrolled. Part 2 will commence following determination of the MTD and RP2D of single-agent GRN-300 in Part 1.
  Overall duration of the study will be approximately 36-48 months, depending on the rate of enrollment and number of subjects enrolled.
  Interventions: Drug: GRN-300; Drug: Paclitaxel

INTERVENTIONS:
Drug: GRN-300 — A salt-inducible kinase (SIK) inhibitor
  Other Names: SIK2/3 Inhibitor
Drug: Paclitaxel — Microtubule inhibitor
  Other Names: Taxane
  Arms: Part 2 (Phase 1b): Single Arm, Open Label (GRN-300 plus paclitaxel)

SUMMARY:
The study consists of two parts based on the administration of single-agent GRN-300 or in combination with paclitaxel.

Part 1 (Phase IA) will test the tolerability of continuous twice a day dosing of oral GRN-300, a salt-inducible kinase inhibitor, with each cycle consisting of 28 days of treatment. The number of administered cycles will depend on the tolerability of each dose level and the severity and occurrence of dose limiting toxicities (DLTs) or adverse events.

Part 2 (Phase IB) will test the tolerability of continuous 28-day cycles of GRN-300 in combination with weekly paclitaxel given 3 of 4 weeks per month (x 3).

Overall duration of the study will be approximately 48 months, depending on the rate of enrollment and number of subjects enrolled.

DETAILED DESCRIPTION:
Part 1: Phase 1A

Primary objectives:

Determination of the maximum tolerated dose (MTD), if applicable, and recommended Phase II dose (RP2D) of GRN-300 in the study population.

To investigate the safety and tolerability of repeated 28-day cycles of oral GRN-300 therapy in subjects with persistent or recurrent, locally non-resectable or metastatic ovarian, fallopian tube, and primary peritoneal cancer or other advanced solid tumors.

Secondary objectives:

To evaluate the pharmacokinetic (PK) profile of GRN-300 after oral administration of a single dose and at steady state.

To estimate the clinical activity of GRN-300 monotherapy by determining the following:

* Overall response rate (ORR) per investigator assessment using RECIST v1.1 defined as the percentage of subjects having a best overall response (BOR) of complete response (CR) or partial response (PR)
* Disease control rate (DCR) per investigator assessment using RECIST v1.1 defined as the percentage of subjects having a BOR of CR, PR, or stable disease (SD) ≥ 4 months (4 cycles, 28 days each).

Part 2: Phase 1B

Primary objectives:

Determination of the RP2D of GRN-300 in combination with weekly paclitaxel given 3 of 4 weeks per month (x 3) in the study population.

To investigate the safety and tolerability of repeated 28-day cycles of daily oral GRN-300 therapy in combination with weekly paclitaxel x 3 in subjects with persistent or recurrent, locally non-resectable or metastatic, ovarian, fallopian tube, and primary peritoneal cancer, where treatment with paclitaxel is appropriate.

Secondary objectives:

To evaluate the PK profile of GRN-300 and paclitaxel following administration of a single dose of each and at steady state.

To estimate the clinical activity of GRN-300 in combination with paclitaxel by determining the following:

* Overall response rate (ORR) per investigator assessment using RECIST v1.1 defined as the percentage of subjects having a best overall response (BOR) of complete response (CR) or partial response (PR)
* DCR per investigator assessment using RECIST v.1.1 defined as the percentage of subjects having a BOR of CR, PR, or SD ≥ 4 months (4 cycles, 28 days each).

Exploratory Translational Objectives for Both Study Parts:

* To estimate progression free survival (PFS) per investigator assessment using RECIST v1.1 for subjects who received continuous GRN-300 and weekly paclitaxel x 3.
* Evaluate exploratory biomarkers of target engagement and treatment response

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Part 1 dose-escalation cohorts: Diagnosis of persistent or recurrent, locally non-resectable or metastatic ovarian, primary peritoneal or fallopian tube epithelial cancer, or advanced solid tumors of any other histology who have progressed on standard therapy and for whom no further effective therapy is available
* Part 1 dose-expansion cohort / Part 2 dose-escalation cohorts / Part 2 dose-expansion cohort: Diagnosis of persistent or recurrent, locally non-resectable or metastatic ovarian, primary peritoneal or fallopian tube epithelial cancer who have progressed on standard therapy and for whom no further effective therapy is available. Patients with advanced solid tumors of any other histology will not be eligible to be enrolled in these cohorts.
* Part 2 dose-escalation cohorts / Part 2 dose-expansion cohort: paclitaxel treatment for the tumor should be indicated
* Histologic or cytologic confirmation of the original tumor by Pathology assessment is required.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension, as defined by RECIST 1.1.
* Prior therapy: Patients must have received at least one prior second-line treatment for persistent, recurrent, locally non-resectable or metastatic disease but may have received any number of prior treatments.
* Any unresolved toxicities from prior therapy should be no greater than NCI-CTCAE v5.0 Grade 1 at screening.
* Patients who are expected to survive a minimum of three months after the first administration of the study drug.
* Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0-1.
* Adequate bone marrow, liver and renal function.

Exclusion Criteria:

* Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug.
* Patients with known hypersensitivity to paclitaxel excluded from Part 2 paclitaxel combination only).
* Use of any cytotoxic chemotherapy or investigational drugs, biologics, or devices within 21 days prior to study enrollment.
* Women who are pregnant or breastfeeding.
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
* Known CNS metastases or leptomeningeal disease.
* Gastrointestinal dysfunction that may affect oral drug absorption (e.g., intermittent or chronic bowel obstruction, short gut, etc.).
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within six months of start of study treatment.
* Other medical co-morbidities that in the investigator's judgment would increase the risks of participation
* QTc >480 msec be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Part 1 (Phase 1A) - Determination of the MTD and the RP2D of GRN-300 single-agent based on evaluation of the DLT in the study population. | 24 months
  • Determination of the recommended Phase II dose (RP2D) of GRN-300 in the study population.
Part 1 (Phase 1A) - Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | 24 months
  • To investigate the safety of repeated 28-day cycles of daily oral GRN-300 therapy in subjects with recurrent or metastatic ovarian, fallopian tube, and primary peritoneal cancer or other advanced solid tumors, based on the number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
Part 2 (Phase 1B) - Determination of the MTD and the RP2D of GRN-300 with paclitaxel based on evaluation of the DLT in the study population | 24 months
  • Determination of the recommended Phase II dose (RP2D) of GRN-300 in combination with weekly paclitaxel in the study population.
Part 2 (Phase 1B) - Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | 24 months
  • To investigate the safety of repeated 28-day cycles of daily oral GRN-300 therapy in combination with weekly paclitaxel x 3 in subjects with recurrent or metastatic ovarian, fallopian tube, and primary peritoneal cancer or other advanced solid tumors, based on the number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Part 1 (Phase 1A) - Determination of GRN-300 monotherapy PK profile (Cmax). | 24 months
  • To evaluate the pharmacokinetic (PK) profile of GRN-300 after oral administration of a single dose and at steady state.
  - Maximum plasma concentration (Cmax)
Part 1 (Phase 1A) - Determination of GRN-300 monotherapy PK profile (tmax). | 24 months
  • To evaluate the pharmacokinetic (PK) profile of GRN-300 after oral administration of a single dose and at steady state.
  - Time to Cmax (tmax)
Part 1 (Phase 1A) - Determination of GRN-300 monotherapy PK profile (t1/2). | 24 months
  • To evaluate the pharmacokinetic (PK) profile of GRN-300 after oral administration of a single dose and at steady state.
  - Terminal half-life (t1/2)
Part 1 (Phase 1A) - Determination of GRN-300 monotherapy PK profile (AUC0-t). | 24 months
  • To evaluate the pharmacokinetic (PK) profile of GRN-300 after oral administration of a single dose and at steady state.
  - Area under the plasma concentration-time curve from zero to the last measurable concentration (AUC0-t)
Part 1 (Phase 1A) - Determination of GRN-300 monotherapy PK profile (AUC0-Inf). | 24 months
  • To evaluate the pharmacokinetic (PK) profile of GRN-300 after oral administration of a single dose and at steady state.
  - Area under the plasma concentration-time curve from zero to infinity (AUC0-Inf)
Part 1 (Phase 1A) - Determination of GRN-300 monotherapy PK profile (CL/F). | 24 months
  • To evaluate the pharmacokinetic (PK) profile of GRN-300 after oral administration of a single dose and at steady state.
  - Apparent oral clearance (CL/F)
Part 1 (Phase 1A) - Determination of GRN-300 monotherapy PK profile (Vz/F). | 24 months
  • To evaluate the pharmacokinetic (PK) profile of GRN-300 after oral administration of a single dose and at steady state.
  - Apparent volume of distribution during terminal distribution phase (Vz/F)
Part 1 (Phase 1A) - Estimation of the clinical activity of single agent GRN-300 (ORR) | 24 months
  • Overall response rate (ORR) per investigator assessment using RECIST v1.1 defined as the percentage of subjects having a best overall response (BOR) of complete response (CR) or partial response (PR)
Part 1 (Phase 1A) - Estimation of the clinical activity of single agent GRN-300 (DCR) | 24 months
  • Disease control rate (DCR) per investigator assessment using RECIST v1.1 defined as the percentage of subjects having a BOR of CR, PR, or stable disease (SD) ≥ 4 months (4 cycles, 28 days each)
Part 2 (Phase 1B) - Determination of GRN-300 plus paclitaxel PK profile (Cmax). | 24 months
  • To evaluate the PK profile of GRN-300 and paclitaxel following administration of a single dose of each and at steady state.
  - Maximum plasma concentration (Cmax)
Part 2 (Phase 1B) - Determination of GRN-300 plus paclitaxel PK profile (tmax). | 24 months
  • To evaluate the PK profile of GRN-300 and paclitaxel following administration of a single dose of each and at steady state.
  - Time to Cmax (tmax)
Part 2 (Phase 1B) - Determination of GRN-300 plus paclitaxel PK profile (t1/2). | 24 months
  • To evaluate the PK profile of GRN-300 and paclitaxel following administration of a single dose of each and at steady state.
  - Terminal half-life (t1/2)
Part 2 (Phase 1B) - Determination of GRN-300 plus paclitaxel PK profile (AUC0-t). | 24 months
  • To evaluate the PK profile of GRN-300 and paclitaxel following administration of a single dose of each and at steady state.
  - Area under the plasma concentration-time curve from zero to the last measurable concentration (AUC0-t)
Part 2 (Phase 1B) - Determination of GRN-300 plus paclitaxel PK profile (AUC0-Inf). | 24 months
  • To evaluate the PK profile of GRN-300 and paclitaxel following administration of a single dose of each and at steady state.
  - Area under the plasma concentration time curve from zero to infinity (AUC0-Inf)
Part 2 (Phase 1B) - Determination of GRN-300 plus paclitaxel PK profile (CL/F). | 24 months
  • To evaluate the PK profile of GRN-300 and paclitaxel following administration of a single dose of each and at steady state.
  - Apparent oral clearance (CL/F)
Part 2 (Phase 1B) - Determination of GRN-300 plus paclitaxel PK profile (Vz/F). | 24 months
  • To evaluate the PK profile of GRN-300 and paclitaxel following administration of a single dose of each and at steady state.
  - Apparent volume of distribution during terminal distribution phase (Vz/F)
Part 2 (Phase 1B) - Estimation of the clinical activity of GRN-300 plus paclitaxel (ORR). | 24 months
  • Overall response rate (ORR) per investigator assessment using RECIST v1.1 defined as the percentage of subjects having a best overall response (BOR) of complete response (CR) or partial response (PR)
Part 2 (Phase 1B) - Estimation of the clinical activity of GRN-300 plus paclitaxel (DCR). | 24 months
  • DCR per investigator assessment using RECIST v.1.1 defined as the percentage of subjects having a BOR of CR, PR, or SD ≥ 4 months (4 cycles, 28 days each)

OTHER OUTCOMES:
Part 1 and 2: progression free survival (PFS) | 48 months
  • To estimate progression free survival (PFS) per investigator assessment using RECIST v1.1 for subjects who received continuous GRN-300 single-agent or in combination with weekly paclitaxel x 3

CONTACTS AND LOCATIONS:
Overall Officials: Siqing Fu, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No